CLINICAL TRIAL: NCT00406120
Title: Validation of a Molecular Test for Predicting Metastasis in Patients With Uveal Melanoma
Brief Title: Validation of a Molecular Prognostic Test for Eye Melanoma
Status: Withdrawn | Type: Observational
Why Stopped: It has come to our attention that the site was not necessary for our research project.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 98-0042-A
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Uveal Neoplasms; Choroid Neoplasms; Iris Neoplasms
Keywords: eye; uvea; iris; choroid; ciliary body; melanoma; iris melanoma; choroidal melanoma; ciliary body melanoma; uveal melanoma; posterior uveal melanoma; prognosis; metastasis; genetic testing; molecular testing; gene expression profiling
MeSH Terms: conditions — Uveal Neoplasms; Choroid Neoplasms; Iris Neoplasms; Melanoma; Uveal Melanoma; Neoplasm Metastasis | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: Fine needle aspiration biopsy

SUMMARY:
Up to half of patients with ocular melanoma (also called iris, choroidal or uveal melanoma) develop metastasis. We have found that certain molecular features of the eye tumor can be detected by gene expression profiling and accurately predict which patients will develop metastasis. This molecular test could eventually allow high risk patients to receive preventative therapy to delay or prevent the development of metastasis. The goal of this study is to prospectively validate the predictive accuracy of the gene expression-based molecular test and compare it to monosomy 3, the most common but potentially less accurate molecular marker for metastasis in ocular melanoma.

DETAILED DESCRIPTION:
We have discovered a gene expression profile derived from primary uveal melanomas that accurately predicts which patients will develop metastasis. Tumors with a class 1 gene expression signature have a very low risk, and those with a class 2 signature have a high risk of metastasis. The molecular test was initially performed on tissue obtained from enucleated eyes using commercial microarray platforms. We are now able to perform the molecular test on fine needle biopsy specimens, and we have developed a customized test that has greater dynamic range and sensitivity than commercial microarray platforms. The goal of this study is to validate the prognostic accuracy of the customized platform by performing the molecular test on primary uveal melanomas obtained from enucleation, local tumor resection or fine needle biopsy. Each sample will be diagnosed as either class 1, class 2 or indeterminate. Outcomes will be collected and the ability of the molecular diagnosis to predict metastasis will be evaluated at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of melanoma of the iris, ciliary body and/or choroid
* treatment to include enucleation, radiotherapy or local tumor resection

Exclusion Criteria:

* evidence of marked tumor necrosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients have uveal melanoma and are being treated wither by enucleation or plaque radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-05 (Estimated); Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Presentation of Primary Tumor to Metastasis | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: J. William Harbour, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Onken MD, Worley LA, Davila RM, Char DH, Harbour JW. Prognostic testing in uveal melanoma by transcriptomic profiling of fine needle biopsy specimens. J Mol Diagn. 2006 Nov;8(5):567-73. doi: 10.2353/jmoldx.2006.060077. PMID 17065425
- [Background] Onken MD, Ehlers JP, Worley LA, Makita J, Yokota Y, Harbour JW. Functional gene expression analysis uncovers phenotypic switch in aggressive uveal melanomas. Cancer Res. 2006 May 1;66(9):4602-9. doi: 10.1158/0008-5472.CAN-05-4196. PMID 16651410
- [Background] Onken MD, Lin AY, Worley LA, Folberg R, Harbour JW. Association between microarray gene expression signature and extravascular matrix patterns in primary uveal melanomas. Am J Ophthalmol. 2005 Oct;140(4):748-9. doi: 10.1016/j.ajo.2005.04.024. PMID 16226537
- [Background] Faulkner-Jones BE, Foster WJ, Harbour JW, Smith ME, Davila RM. Fine needle aspiration biopsy with adjunct immunohistochemistry in intraocular tumor management. Acta Cytol. 2005 May-Jun;49(3):297-308. doi: 10.1159/000326153. PMID 15966293
- [Background] Onken MD, Worley LA, Ehlers JP, Harbour JW. Gene expression profiling in uveal melanoma reveals two molecular classes and predicts metastatic death. Cancer Res. 2004 Oct 15;64(20):7205-9. doi: 10.1158/0008-5472.CAN-04-1750. PMID 15492234